CLINICAL TRIAL: NCT02719197
Title: Single-center, Double-blind, Placebo-controlled, Randomized, Single-ascending Dose Study to Investigate the Tolerability, Safety, Pharmacokinetics (Including Food Effect), and Pharmacodynamics of an Oral Drug for Neurological Disorders in Healthy Male Subjects
Brief Title: First-in-man Study of Single Ascending Dose of a New Drug for Neurological Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AC-083-101; 2015-005012-15 (EudraCT Number)
Record Dates: First submitted 2016-03-14; First posted 2016-03-25 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AC-083, Single Ascending Dose (Experimental): AC-083 administered at different single dose levels in a sequential manner, and in a maximum of 9 dose levels starting from 1 mg (number of cohorts and dose levels will depend on the safety and pharmacokinetic results of the previous cohort). Each dose level will be investigated in a new group of 8 healthy male subjects (6 on active drug and 2 on placebo)
  Interventions: Drug: AC-083
- Placebo, Single Ascending Dose (Placebo Comparator): Matched placebo administered as single ascending doses in parallel to AC-083
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AC-083 — Hard gelatin capsules for oral administration formulated at a strengths of 1, 10 and 100 mg
  Arms: AC-083, Single Ascending Dose
Drug: Placebo — Placebo capsules matching AC-083 capsules
  Arms: Placebo, Single Ascending Dose

SUMMARY:
The primary purpose of this first-in-man study is to investigate whether a new drug for neurological disorders is safe and well-tolerated when administered orally to healthy male adults

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy on the basis of physical examination, electrocardiogram and laboratory tests.
* A subject who has a female partner of childbearing potential or a pregnant partner agrees to use a condom in combination with spermicide or a condom, respectively, from screening, during the entire study, and for at least 3 months after (the last) study drug intake
* Body mass index (BMI) of 18.0 to 29.9 kg/m2 (inclusive) at screening and Day -1.
* Systolic blood pressure (SBP) 100-140 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and pulse rate 50-90 bpm (inclusive), measured after 5 min in the supine position at screening and at Day -1.

Exclusion Criteria:

* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study treatment
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions
* Any cardiac condition or illness with a potential to increase the cardiac risk of the subject based on medical history, physical examination, or electrocardiogram (ECG) evaluations
* Any circumstances or conditions, which, in the opinion of the Investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From baseline to end of study (EOS) (up to Day 12)
  Treatment-emergent AEs and treatment emergent serious AEs
Changes from baseline in supine blood pressure | From baseline to EOS (up to Day 12)
  Supine blood pressure (mmHg)
Changes from baseline in electrocardiogram (ECG) variables | From baseline to EOS (up to Day 12)
  ECG variables are to be recorded at rest using a standard 12-lead ECG
Changes from baseline in pulse rate | From baseline to EOS (up to Day 12)
  Pulse rate (bpm)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) following single oral ascending doses | From pre-dose on Day 1 to up to Day 12
  Cmax is derived from the observed plasma concentration-time curves
Time to reach Cmax (tmax) following single oral ascending doses | From pre-dose on Day 1 to up to Day 12
  Tmax is derived from the observed plasma concentration-time curves
Terminal half-life [t(1/2)] following single oral ascending doses | From pre-dose on Day 1 to up to Day 12
Area under the plasma concentration-time curve (AUC) following single oral ascending doses | From pre-dose on Day 1 to up to Day 12
  AUC is defined for the time intervals from zero to time t of the last measured concentration above the limit of quantification, from zero to infinity and from zero to 24 h after study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Investigator Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No